CLINICAL TRIAL: NCT06304233
Title: The Protein Disrupted in Schizophrenia 1 (DISC1) as a Novel Biomarker for Cardiac Disease - The Link Between DISC1 and Cardiac Function in Patients With Schizophrenia
Brief Title: The Protein Disrupted in Schizophrenia 1 (DISC1) as a Novel Biomarker for Cardiac Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 606103
Record Dates: First submitted 2023-12-11; First posted 2024-03-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Heart Diseases; Heart; Functional Disturbance; Schizophrenia
Keywords: Disrupted in Schizophrenia 1; DISC1; Cardiac Biomarker
MeSH Terms: conditions — Heart Diseases; Schizophrenia | interventions — Echocardiography; Caves; Electrocardiography; Electrocardiography, Ambulatory; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, whole blood, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnosed with Schizophrenia: Patients with a ICD-10 diagnosis of Schizophrenia will undergo investigations to assess cardiac function, cardiovascular disease risk factors and DISC1 mRNA expression. Participants eligible for MRI will be invited to undergo cardiac MRI in addition to echocardiography.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Cardiac Magnetic Resonance Imaging; Diagnostic Test: Electrocardiography; Other: Blood sampling
- No mental health diagnosis: Participants without a mental health diagnosis will be randomly selected from an existing population registered in the HUNT data and biobank for whom, echocardiographic data and biological samples are available.Those enrolled as controls will be invited to participate in the cardiac MRI portion of the study.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Cardiac Magnetic Resonance Imaging; Diagnostic Test: Electrocardiography; Other: Blood sampling

INTERVENTIONS:
Diagnostic Test: Echocardiography — ultrasound assessment of heart structure, volume and function
  Other Names: Echo
Diagnostic Test: Cardiac Magnetic Resonance Imaging — MRI assessment of heart structure, volume, function and tissue characteristics
  Other Names: Cardiac MRI; CMRI
Diagnostic Test: Electrocardiography — Assessment of cardiac rhythm and electrical activity
  Other Names: Holter; ECG
Other: Blood sampling — To measure DISC1 mRNA expression and other potential biomarkers

SUMMARY:
To study the association between DISC1 RNA expression levels and cardiac function in patients with schizophrenia.

DETAILED DESCRIPTION:
Potential participants interested in the study will be screened for eligibility. Those who meet the eligibility criteria will be informed about the study, the expected investigations and its potential risks. All participants giving written informed consent will be enrolled into the study. Participants will be interviewed, given questionnaires, have blood and/or skin samples and clinical parameters taken. Cardiac function parameters will be measured using electrocardiography, echocardiography and magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ICD-10 schizophrenia, schizotypal or delusional disorders (F20 to F29)
* Both inpatient and outpatient
* Capable of giving informed consent

Exclusion Criteria:

* Current or previous diagnosis of cancer
* Current or previous treatment with chemotherapy
* Current pregnancy
* Mothers less than 6 months post-partum

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort with schizophrenia will be recruited from outpatient and inpatient population from a single centre.
  The cohort without mental health diagnosis will be selected from an existing population registered in the HUNT data and biobank and be matched for age (± 2 years) and sex of the patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2038-06 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) measured by 2D Echocardiography | Baseline
  Left ventricular ejection fraction, LVEF will be reported in percentage (%) and obtained using Simpson's biplane method from 2D echocardiography.
Left Ventricular Ejection Fraction (LVEF) measured by 3D Echocardiography | Baseline
  Left ventricular ejection fraction, LVEF will be reported in percentage (%) and obtained using 3D echocardiography
DISC1 mRNA quantification | Baseline
  Measured from blood samples and reported as fold change
Levels of high sensitive-CRP | Baseline
  Levels of HS-CRP mg/L
Levels of CK-MB | Baseline
  Levels of CK-MB is reported in µg/L
Levels of Troponin T | Baseline
  Levels of Troponin T is reported in ng/L
Levels of Troponin I | Baseline
  Levels of Troponin I is reported in ng/L
Normalized Left Ventricular End-Diastolic Volume (LV EDV), echocardiographic parameter | Baseline
  LV EDV in milliliters (mL) will be normalized against body surface area (BSA) in m^2 to report LV EDV normalized by BSA in mL/m^2.
Normalized Right Ventricular End-Diastolic Volume (RV EDV), echocardiographic parameter | Baseline
  RV EDV in mL will be normalized against body surface area (BSA) in m^2 to report RV EDV normalized by BSA in mL/m^2.
Normalized left Ventricular End-Systolic Volume (LV ESV), echocardiographic parameter | Baseline
  LV ESV in mL will be normalized against body surface area (BSA) in m^2 to report LV ESV normalized by BSA in mL/m^2.
Normalized Right Ventricular End-Systolic Volume (RV ESV), echocardiographic parameter | Baseline
  RV ESV in mL will be normalized against body surface area (BSA) in m^2 to report RV ESV normalized by BSA in mL/m^2.
Left ventricular mass measured by echocardiography | Baseline
  Left ventricular mass in grams (g) will be normalized against BSA in m^2 and reported as g/m ^2
Left ventricular septal thickness, left ventricular posterior wall thickness and right ventricular wall thickness measured by echocardiography | Baseline
  Left ventricular septal thickness, left ventricular posterior wall thickness and right ventricular wall thickness will be reported in centimeters (cm)
Fractional shortening measured by echocardiography | Baseline
  Fractional shortening will be reported as a percentage (%)
Global longitudinal strain (GLS), echocardiographic parameter | Baseline
  GLS(%) = (MLs - MLd)/MLd, where MLs is myocardial length at end-systole and MLd is the myocardial length at end-diastole. GLS will be reported in precentage (%)
TAPSE echocardiographic parameter of right ventricular longitudinal systolic function | baseline
  TAPSE will be reported in millimeters (mm)
Echocardiographic parameter MPI, Myocardial performance index | Baseline
  MPI is a unitless index derived from the sum of the isovolumic relaxation time (IVRT) and the isovolumic contraction time (IVCT) in milliseconds (ms) divided by the ejection time interval in (ms).
Echocardiographic parameter Mitral E/A ratio | Baseline
  Mitral E/A ratio is derived from the ratio of the E wave velocity to the A wave velocity
Echocardiography parameter of peak E velocity | Baseline
  peak E velocity is reported in cm/s
Echocardiography parameter of E wave deceleration time | Baseline
  E wave deceleration time is reported in milliseconds (ms)
Echocardiography parameter of ratio of E/e' | Baseline
  The E/e' ratio is derived from the E wave velocity to the e' velocity
Echocardiographic parameters septal e' and lateral e' velocities | Baseline
  Septal e' and lateral e' velocities are reported as cm/s
Echocardiographic parameter LAVI, left atrial volume indexed | Baseline
  LAVI is reported in mL/m^2 and is the volume (mL) of the left atrium indexed against the BSA in m^2.
Echocardiographic parameter TRpV, Tricuspid Regurgitation peak Velocity | Baseline
  TRpV is reported in m/s
Echocardiographic parameter, S wave velocity | Baseline
  S wave velocity is the peak systolic velocity of the tricuspid annulus and is reported in cm/s
Echocardiographic parameter, Indexed LV and RV stroke volumes | Baseline
  Indexed LV stroke volume and Indexed RV stroke volume will be reported in mL/m^2 by by indexing the volumes (mL) to BSA (m^2)
Levels of NT-proBNP | Baseline
  Levels of NT-proBNP from blood samples will be reported in ng/L
Levels of IGF1 | Baseline
  Levels of IGF1 from blood samples will be reported in nmol/L
Levels of ANP | Baseline
  Levels of ANP from blood samples will be reported in pg/mL
Levels of BDNF, brain derived neurotrophic factor | Baseline
  Levels of BDNF from blood samples will be reported in ng/mL
Levels of Tumor Necrosis Factor alpha | Baseline
  Levels of Tumor Necrosis Factor alpha from blood samples will be reported in pg/mL
Levels of Transforming Growth Factor Beta | Baseline
  Levels of Transforming Growth Factor Beta from blood samples will be reported in ng/mL
Levels of cardiac Myosin-Binding Protein C | Baseline
  Levels of cardiac Myosin-Binding Protein C from blood samples will be reported in ng/L
Interleukin levels | Baseline
  Interleukin levels from blood sample will be reported as pg/mL

SECONDARY OUTCOMES:
native T1 time, cardiac MRI | Baseline
  native myocardial T1 relaxation time is reported in milliseconds (ms)
Indexed LV and RV end-diastolic, end-systolic and stroke volumes, cardiac MRI | Baseline
  Indexed LV and RV end-diastolic, end-systolic and stroke volumes will be reported in mL/m^2, by indexing the volumes (mL) to BSA (m^2)
Indexed LV mass, cardiac MRI | Baseline
  Indexed LV mass will be reported in g/m^2 by indexing mass (g) to BSA (m^2)
LV Ejection Fraction, cardiac MRI | Baseline
  LVEF will be reported in percent (%)
ECG corrected QT interval | Baseline
  corrected QT interval will be reported in milliseconds (ms)
Number of participants with and abnormal ECG | Baseline
  Number of participants with an abnormal ECG will be reported in %
Number of participants with abnormal liver function | Baseline
  Number of participants with abnormal liver function will be reported as %
Number of participants with abnormal kidney function | Baseline
  Number of participants with abnormal kidney function will be reported as %
Number of participants with abnormal thyroid function | Baseline
  Number of participants with abnormal thyroid function will be reported as %
Number of participants with low Vitamin D levels | Baseline
  Number of participants with low Vitamin D levels will be reported as %
Incidence of cardiovascular disease or mortality as registered in a health registry on follow up | Within 15 years from start of study
  Extraction of information from the cardiovascular disease registry and deaths registry between 10 - 15 years from the start of the study to determine incidence of cardiovascular disease outcomes for the study cohort
Triglyceride levels | Baseline
  Triglyceride will be reported in mmol/L
High-density lipoprotein, HDL-cholesterol levels | Baseline
  HDL-cholesterol levels will be reported in mmol/L
Low-density lipoprotein, LDL-cholesterol levels | Baseline
  LDL-cholesterol levels will be reported in mmol/L
Fasting glucose levels | Baseline
  Fasting glucose levels will be reported in mmol/L
Glycated Hemoglobin (HbA1c) levels | Baseline
  HbA1C will be reported in mmol/mol
Heart rate measured on ECG | Baseline
  Heart rate measured on 12 lead ECG will be reported in beats per minute.
Systolic Blood Pressure | Baseline
  Systolic Blood Pressure will be reported as mmHg
Diastolic Blood Pressure | Baseline
  Diastolic Blood Pressure will be reported as mmHg
Lipoprotein a | Baseline
  Lipoprotein a levels will be reported in mg/L
Magnesium levels | Baseline
  Magnesium levels will be reported as mmol/L
Calcium levels | Baseline
  Calcium levels will be reported as mmol/L
Sodium levels | Baseline
  Sodium levels will be reported as mmol/L
Potassium levels | Baseline
  Potassium levels will be reported as mmol/L

OTHER OUTCOMES:
Alcohol intake at baseline using The Alcohol Use Disorders Identification Test Consumption (AUDIT-C) questionnaire | Baseline
  The AUDIT-C is a validated 3-item questionnaire for identification of alcohol misuse. Each item has 5 possible responses, each scored from 0 to 4 points. Possible scores range from 0 to 12. The score cut-off for alcohol misuse is 4 points in men and 3 points in women
Average length of inpatient stay for schizophrenia related admissions | Baseline
  The average length of inpatient stays will be reported as number of days and derived from the total number of days spent admitted over the total number of admissions.
Need of Care based on number of total hospital admission for schizophrenia | Baseline
  Number of hospital admissions
Severity scoring of psychiatric symptoms using Clinical Global Impressions (CGI) Scale - Severity | Baseline
  CGI for severity is a validated scale used to assess psychiatric illness severity by a clinician. Possible scores range from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients)
Schizophrenia symptom severity as scored on the Positive and Negative Syndrome Scale (PANSS) | Baseline
  PANSS/SCI-PANSS are validated clinician administered scale used to measure symptom severity in schizophrenia and consists of 30 items divided into 3 subscales: Positive Scale, Negative Scale and the General Pathology Scale. Each subscale can be scored from 1 (absent) to 7 (extreme). Possible scores for the Positive and Negative scales range from 7 - 49, and for the General Psychopathology Scale range from 16 - 112. The further developed SCI-PANSS (structured clinical interview - for the Positive and Negative Syndrome Scale).
Duration of schizophrenia | Baseline
  Duration of schizophrenia as determined from self reported year of first episode of diagnosis/ or from date of diagnosis
Length of treatment with an antipsychotic medication | Baseline
  The length of treatment with an antipsychotic medication will be reported in years
Antipsychotic dosage in daily equivalent dosage of chlorpromazine | Baseline
  Antipsychotic dosages will also be converted to daily equivalent dosage of chlorpromazine for comparison across different medication will be reported in mg/day
Smoking status | Baseline
  Number of participants who smoke will be reported in percent (%)
Waist Hip Ratio | Baseline
  Waist Hip measurements will be reported as a ratio
Body Mass Index | Baseline
  Body Mass Index, BMI will be derived from participants weight and height and reported as kg/m^2
Body fat percent | Baseline
  Body fat percent from body composition analysis will be reported in %
Physical Activity | Baseline
  Baseline physical activity measured using the International Physical Activity Questionnaire (IPAQ) The IPAQ is validated in schizophrenia populations and the IPAQ has been validated in Norwegian populations. It is a self reported scoring system assessing physical activity over the last seven days. Physical activity can be then represented in minutes/week or MET-minutes/week.
Body muscle composition | Baseline
  Body muscle mass will be reported in kg
Smoking history | Baseline
  Smoking will be quantified and reported as pack/years
Age of participant | Baseline
  Age of participant will be reported in years
Gender of participant | Baseline
  Gender of participant will be reported as male or female

CONTACTS AND LOCATIONS:
Overall Officials: Morten A Høydal, PhD, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Norwegian University of Science and Technology, Trondheim
  - St Olavs Hospital, Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the study, after deidentification can be shared.
Supporting Information: Study Protocol
Time Frame: During the whole project period up to 15 years.
Access Criteria: For cooperative research and publication within Norway, the EU and the US, for purposes inline with those in the Study protocol.